CLINICAL TRIAL: NCT04940559
Title: A Phase 1 Study To Determine The Relative Bioavailability Of ACH-0144471 After Administration Of A Tablet Or Softgel Capsule Versus A Liquid Filled Capsule In Healthy Volunteers
Brief Title: Study of Different Forms of Danicopan (Tablet, Softgel Capsule, Liquid-filled Capsule) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Achillion, a wholly owned subsidiary of Alexion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ACH471-006; ACTRN12616001017415 (Registry Identifier: ANZCTR)
Record Dates: First submitted 2021-06-21; First posted 2021-06-25 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Healthy
Keywords: Danicopan; ALXN2040; ACH-0144471; Relative Bioavailability; LFC; Tablet; Softgel Capsule; Food Effect; Pharmacokinetics; Factor D Inhibitor; Safety
MeSH Terms: interventions — danicopan; rhoA GTP-Binding Protein

STUDY DESIGN:
Intervention Model Description: Group 1 followed a 3-treatment, 3-period crossover study design. Group 2 followed a 2-treatment, 2-period crossover study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group 1: Sequence 1 (Experimental): Participants received danicopan once each period as a single dose under fasted or fed (medium-fat meal) conditions as follows:
  Period 1: Danicopan as an LFC under fasted conditions. Period 2: Danicopan as a tablet under fed (medium-fat meal) conditions. Period 3: Danicopan as a tablet under fasted conditions. There was a washout period of at least 4 days (96 hours) between each danicopan dosing.
  Interventions: Drug: Danicopan - Tablet; Drug: Danicopan - LFC
- Group 1: Sequence 2 (Experimental): Participants received danicopan once each period as a single dose under fasted or fed (medium-fat meal) conditions as follows:
  Period 1: Danicopan as a tablet under fed (medium-fat meal) conditions. Period 2: Danicopan as a tablet under fasted conditions. Period 3: Danicopan as an LFC under fasted conditions. There was a washout period of at least 4 days (96 hours) between each danicopan dosing.
  Interventions: Drug: Danicopan - Tablet; Drug: Danicopan - LFC
- Group 1: Sequence 3 (Experimental): Participants received danicopan once each period as a single dose under fasted or fed (medium-fat meal) conditions as follows:
  Period 1: Danicopan as a tablet under fasted conditions. Period 2: Danicopan as an LFC under fasted conditions. Period 3: Danicopan as a tablet under fed (medium-fat meal) conditions. There was a washout period of at least 4 days (96 hours) between each danicopan dosing.
  Interventions: Drug: Danicopan - Tablet; Drug: Danicopan - LFC
- Group 2: Sequence 1 (Experimental): Participants received danicopan once each period as a single dose under fasted conditions as follows:
  Period 1: Danicopan as an LFC under fasted conditions. Period 2: Danicopan as a softgel capsule under fasted conditions. There was a washout period of at least 4 days (96 hours) between each danicopan dosing.
  Interventions: Drug: Danicopan - Softgel; Drug: Danicopan - LFC
- Group 2: Sequence 2 (Experimental): Participants received danicopan once each period as a single dose under fasted conditions as follows:
  Period 1: Danicopan as a softgel capsule under fasted conditions. Period 2: Danicopan as an LFC under fasted conditions. There was a washout period of at least 4 days (96 hours) between each danicopan dosing.
  Interventions: Drug: Danicopan - Softgel; Drug: Danicopan - LFC

INTERVENTIONS:
Drug: Danicopan - Tablet — Oral tablet.
  Other Names: ALXN2040; ACH-0144471 (formerly); ACH-4471; ACH4471; 4471
  Arms: Group 1: Sequence 1; Group 1: Sequence 2; Group 1: Sequence 3
Drug: Danicopan - Softgel — Oral softgel capsule.
  Other Names: ALXN2040; ACH-0144471 (formerly); ACH-4471; ACH4471; 4471
  Arms: Group 2: Sequence 1; Group 2: Sequence 2
Drug: Danicopan - LFC — Oral LFC.
  Other Names: ALXN2040; ACH-0144471 (formerly); ACH-4471; ACH4471; 4471

SUMMARY:
This was a randomized, crossover, open-label study to assess the relative bioavailability, pharmacokinetics (PK), and safety of three different formulations of danicopan (tablet, softgel capsule, liquid-filled capsule [LFC]) in healthy participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy was defined as having no clinically relevant abnormalities identified by a detailed medical history, physical examination, blood pressure and heart rate measurements, 12-lead electrocardiogram, and clinical laboratory tests.
* Had a body mass index of 18 to 30 kilograms(kg)/meter squared with a minimum body weight of 50 kg.

Key Exclusion Criteria:

* History or clinically relevant evidence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease.
* History of procedures that could alter absorption of orally administered drugs.
* Body temperature ≥ 38°Celsius on Day -1 or Day 1 predose; history of febrile illness within 7 days prior to study drug administration.
* Positive alcohol and/or drug screen at Screening or Day -1; current tobacco/nicotine user.
* Participation in a clinical study within 30 days prior to study drug administration.
* Clinically significant laboratory abnormalities at Screening or Day -1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2016-08-02 (Actual); Primary Completion 2016-10-05 (Actual); Study Completion 2016-10-05 (Actual)

PRIMARY OUTCOMES:
PK: Maximum Plasma Concentration (Cmax) Of Danicopan After Treatment With Each Of The Three Formulations | Up to 96 hours postdose
PK: Time To Reach The Maximum Plasma Concentration (Tmax) Of Danicopan After Treatment With Each Of The Three Formulations | Up to 96 hours postdose
PK: Area Under The Plasma Concentration-time Curve Extrapolated To Infinity (AUC0-Inf) Of Danicopan After Treatment With Each Of The Three Formulations | Up to 96 hours postdose

SECONDARY OUTCOMES:
PK: Cmax Of Danicopan After Treatment With The Tablet Under Fed And Fasted Conditions | Up to 96 hours postdose
PK: Tmax Of Danicopan After Treatment With The Tablet Under Fed And Fasted Conditions | Up to 96 hours postdose
PK: AUC0-inf Of Danicopan After Treatment With The Tablet Under Fed And Fasted Conditions | Up to 96 hours postdose
Incidence Of Serious Adverse Events, Grade 3 Or 4 Adverse Events (AEs), And AEs Leading To Discontinuation | Day 1 through Day 39

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Site, Auckland, New Zealand